CLINICAL TRIAL: NCT04214678
Title: DeFect cLOsure After Colonic ESD With underwaTer Technique Versus Conventional Clip : a Randomized Controlled Trial
Brief Title: DeFect cLOsure After Colonic ESD With underwaTer Technique
Acronym: FLOAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Hon Chi Yip, Associate Consultant, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE 2019.558
Record Dates: First submitted 2019-12-28; First posted 2020-01-02 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Colonic Polyp
Keywords: Endosocpic submucosal dissection; Underwater clip closure
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Underwater clip closure (Experimental): The post-resection defect is closed using endoscopic clips with underwater technique
  Interventions: Procedure: Underwater clip closure
- Conventional clip closure (Active Comparator): The post-resection defect is closed using endoscopic clips with conventional gas insufflation (CO2)
  Interventions: Procedure: Conventional clip closure

INTERVENTIONS:
Procedure: Underwater clip closure — Closure of post-resection defect with endoscopic clips by underwater technique
  Arms: Underwater clip closure
Procedure: Conventional clip closure — Closure of post-resection defect with endoscopic clip by conventional technique
  Arms: Conventional clip closure

SUMMARY:
This is a single centre randomised controlled study comparing underwater clip closure versus conventional gas insufflation clip closure of post-resection defect in patients undergoing colonic endoscopic resection. The investigators hypothesize that underwater clip closure would be faster than conventional closure under gas insufflation.

DETAILED DESCRIPTION:
Endoscopic submucosal dissection (ESD) is a minimally invasive technique that has been increasingly applied to superficial colorectal tumours over the past two decades (1, 2). Although serious complications with this procedure are uncommon, both significant delayed haemorrhage (1-2%) and perforation (4-6%) are recognised complications (3). Although perforation is generally recognised and treated at time of endoscopy, delayed bleeding often requires repeat readmission and endoscopy for haemorrhage control. There is growing evidence to support prophylactic clip closure of mucosal defects to reduce incidences of delayed haemorrhage.

Prophylactic clip closure of mucosal defects (≥20mm) after colonic ESD is supported by large retrospective case series. In a series of 524 lesions in 463 patients, Liaquat et al. (2013) reported prophylactic clipping of resection sites to close mucosal defects versus non-closure, reduced delayed haemorrhage (9.7% vs 1.8%) (4). Ogiyama et al. (2018) reported similar findings in a series of 156 lesions (0% vs 8.2%, p=0.008) (5).

Prophylactic defect closure also has a theoretical benefit in reducing delayed perforation from unrecognised muscular breach during dissection. Though it is recognised that there is a paucity of evidence to support mucosal apposition in reducing delayed perforation rates (~0.2%) (3). This is likely due to the underpowered published studies and a very low event rate.

For these reasons, it has been routine practice of many endoscopists for clip closure of mucosal defects after endoscopic resection of large colorectal neoplasia. However, this technique remains technically challenging within the narrow colonic space and at times may not be feasible. The 'underwater closure technique' in mucosal defect closure of colonic and duodenal endoscopic resections has promising early results. Compared to conventional CO2 insufflation clip placement, at the time of mucosal closure this technique applies luminal water infusion to 'float' the resection borders and downsize the target. Early experience suggests this technique facilitates easier apposition of resection borders and complete closure. There are currently no randomized trials comparing these clip closure techniques.

The aim of the study is to evaluate whether prophylactic underwater closure technique facilitates easier ESD mucosal defect closure compared to conventional clip closure.

This is a single centre prospective randomized controlled trial. Consecutive patients undergoing endoscopic resection for colonic lesions would be recruited. Participants would be randomized to receive prophylactic conventional clip closure versus underwater technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective endoscopic resection
* Colorectal superficial neoplasm with a resultant mucosal defect of ≥20mm
* Age >18 years old

Exclusion Criteria:

* Patients on anticoagulation (Warfarin or other direct oral anticoagulants)
* Muscular perforation during the endoscopic resection
* Incomplete endoscopic resection
* Lesions arising from surgical anastomotic site
* Marked electrolyte abnormalities
* Other cases deemed by the examining physician as unsuitable for safe treatment
* Patients who refused to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Time required to complete clip closure of mucosal defect | Within 1 hour
  o Defined as the time from completion of prophylactic coagulation till the final clip application (min)

SECONDARY OUTCOMES:
Technical success of complete closure of defect (%) | Within 1 hour
Total time for endoscopic procedure (min) | Within 1 hour
Number of endoscopic clip used for closure | Within 1 hour
Rate of Haemorrhage | 30 days
  Post-procedural per rectal bleeding that requires intervention or blood product transfusion
Rate of Perforation | 30 days
  Abdominal pain with radiological evidence of intra-abdominal free gas suggesting perforation
Rate of Post-polypectomy electrocoagulation syndrome | 30 days
  Abdominal pain without radiological evidence of intra-abdominal free gas to suggest perforation
Rate of Any other adverse event related to the procedure | 30 days
  Other adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Hon Chi Yip, MBChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No